CLINICAL TRIAL: NCT03138941
Title: Validation of the Lupus Low Disease Activity State (LLDAS) in the Asia Pacific Region
Acronym: APLCLLDAS
Status: Recruiting | Type: Observational
Sponsor: Monash University (Other)
Collaborators: Flinders Medical Centre, Adelaide, AUSTRALIA (Unknown); St. Vincent's Hospital, Melbourne, AUSTRALIA (Unknown); Royal Adelaide Hospital, Adelaide, AUSTRALIA (Unknown); University of New South Wales, Sydney, AUSTRALIA (Unknown); People's Hospital, Peking University Health Science Center, Beijing, CHINA (Unknown); Peking University First Hospital, Beijing, CHINA (Unknown); The University of Hong Kong (Other); University of Padjadjaran, Bandung, INDONESIA (Unknown); Tokyo Women's Medical University, JAPAN (Unknown); University of Occupational and Environmental Health, JAPAN (Unknown); Keio University, JAPAN (Unknown); Hanyang University Hospital for Rheumatic Diseases, REPUBLIC OF KOREA (Unknown); University of Santo Tomas Hospital, Philippines (Other); National University Hospital, Singapore (Other); Tan Tock Seng Hospital (Other); Chang Gung Memorial Hospital (Other); Taichung Veterans General Hospital (Other); Chiang Mai University Hospital, THAILAND (Unknown); Middlemore Hospital, New Zealand (Other); North Shore Hospital, Auckland, NEW ZEALAND (Unknown); Auckland District Health Board, Auckland, NEW ZEALAND (Unknown); Teaching Hospital Kandy, SRI LANKA (Unknown); University of the Philippines, Philippines (Unknown)
Responsible Party: Sponsor
Other Study IDs: APLC LLDAS Study
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lupus Low Disease Activity State (LLDAS) study is an international, multi-centre prospective study, developed by the Asia Pacific Lupus Collaboration (APLC) to investigate whether the attainment of LLDAS is associated with improved outcomes in patients with Systemic Lupus Erythematosus (SLE).

SLE, or lupus, is the archetypal multisystem autoimmune disease, with an estimated incidence of 5-50 cases per 100,000 people. Patients with SLE, usually young women, suffer a marked loss of life expectancy, and severe morbidity, due to a heterogeneous range of clinical manifestations caused by autoimmune-mediated inflammation of multiple organs. The most severe manifestations of SLE are the accrual of irreversible organ damage, especially renal and central nervous system (CNS) involvement. As there is no effective targeted monotherapy for SLE, patients also suffer severe toxicity from the use of glucocorticoids and broad-spectrum immunosuppressive therapies. Despite combination therapy with current drugs, many studies show that the majority of patients suffer inadequate disease control and inexorably accrue permanent organ damage over time.

The diversity of clinical features of active SLE has made quantification of disease activity problematic. Although there are a number of published systems in use to measure SLE disease activity, there are widely acknowledged problems with these instruments. Published definitions of remission are so stringent that they are met by less than 5% of patients. This lead to the realisation that rather than lupus remission, a lupus low disease activity state target may be more feasible, and that patients with low disease activity are more homogeneous than patients with active disease. Thus, the development of a definition of lupus low disease activity, which is feasible and has face validity, escapes the complexity of attempts to quantify heterogeneous states of active disease.

In this study, the investigators will prospectively collect longitudinal data on consecutive SLE patients at each centre to evaluate the LLDAS definition. Protection from organ damage accrual as the primary endpoint.

DETAILED DESCRIPTION:
In this study, patients with SLE will be followed for ~ 5 years. Regular recordings of the data needed to score LLDAS (disease activity and treatment domains, see Franklyn L et al, Ann Rheum Dis 2016) will be collected, as well as annual recording of lupus-related damage using the SLICC_ACR Damage Index (SDI) and quality of life using the Short Form 36 version 2 (SF36v2).

At conclusion of primary data collection, the associate of LLDAS attainment, or sustained attainment, with protection from organ damage accrual will be ascertained.

ELIGIBILITY:
Inclusion Criteria:

* All patients have to meet either the 1997 American College of Rheumatology (ACR) Modified Classification Criteria for SLE, with at least four of the 11 items; or alternatively, fulfil the Systemic Lupus International Collaborating Clinics (SLICC) 2012 Classification Criteria, with at least four of the 17 items (at least one clinical and one immunological criterion) or with lupus nephritis in the presence of at least one immunological criteria. Patients can be either newly diagnosed or longstanding lupus patients.

All patients must be over the age of 18 and competent to provide written consent.

Exclusion Criteria:

* Patients less than 18 years of age and patients who are unable to consent are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult SLE patients with confirmed lupus
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
SLICC-ACR Damage Index | Approximately 5-10 years
  Organ damage accrual

SECONDARY OUTCOMES:
SFv2-36 | Approximately 5-10 years
  Quality of Life
Mortality | Approximately 5-10 years
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Eric Morand, Study Chair — Monash University
Locations (20):
- Australia (4):
  - Rheumatology Unit, Royal Adelaide Hospital, Adelaide, South Australia
  - Department of Rheumatology, Flinders Medical Centre, Adelaide, South Australia
  - School of Clinical Sciences at Monash Health, Faculty of Medicine, Nursing & Health Sciences, Clayton, Victoria
  - Department of Rheumatology, St Vincent's Hospital (Melbourne), Fitzroy, Victoria
- China (2):
  - Department of Rheumatology and Immunology, People's Hospital Peking University Health Science Center, Beijing, Western District
  - Rheumatology and Immunology department, Peking University First Hospital, Beijing, Xicheng District
- Division of Rheumatology & Clinical Immunology, Department of Medicine, Queen Mary Hospital, the University of Hong Kong, Pok Fu Lam, Hong Kong
- Division of Rheumatology, Department of Internal Medicine, Faculty of Medicine, Padjadjaran University/ Hasan Sadikin General Hospital, Bandung, West Java, Indonesia
- Japan (3):
  - The First Department of Internal Medicine, School of Medicine, University of Occupational and Environmental Health, Kitakyushu
  - Division of Rheumatology, Department of Internal Medicine, School of Medicine, Keio University, Tokyo
  - Institute of Rheumatology, Tokyo Women's Medical University, Tokyo
- Philippines (2):
  - Joint and Bone Center, University of Santo Tomas Hospital, Manila
  - University of the Philippines, Quezon City
- Singapore (2):
  - Rheumatology Division, University Medical Cluster, National University Hospital, Singapore
  - Department of Rheumatology, Allergy & Immunology, Tan Tock Seng Hospital, Tan Tock Seng
- Department of Rheumatology, Hanyang University Hospital for Rheumatic Diseases, Seoul, South Korea
- Division of Nephrology, Teaching Hospital Kandy, Sri Lanka, Kandy, Sri Lanka
- Taiwan (2):
  - Department of Rheumatology, Allergy and Immunology Chang Gung Memorial Hospital Chang Gung University, Guishan, Taoyuan County
  - Division of Allergy, Immunology and Rheumatology, Taichung Veterans General Hospital, Taichung
- Division of Rheumatology, Department of Internal Medicine, Faculty of Medicine, Chiang Mai University Hospital, Chiang Mai, Muang District, Thailand

IPD SHARING:
Plan to Share IPD: No
Patient data collected and collated by the Asia Pacific Lupus Collaboration (APLC) is guided by strict protocols and procedures to ensure that privacy and other ethical principles are maintained at all times. Data sharing will strictly follows the APLC Data Access Policy. Under no circumstances will individual subject data be made available to any third parties.

REFERENCES:
- [Background] Golder V, Huq M, Franklyn K, Calderone A, Lateef A, Lau CS, Lee ALH, Navarra STV, Godfrey T, Oon S, Hoi AYB, Morand EF, Nikpour M. Does expert opinion match the operational definition of the Lupus Low Disease Activity State (LLDAS)? A case-based construct validity study. Semin Arthritis Rheum. 2017 Jun;46(6):798-803. doi: 10.1016/j.semarthrit.2017.01.007. Epub 2017 Jan 18. PMID 28216192
- [Background] Golder V, Kandane-Rathnayake R, Hoi AY, Huq M, Louthrenoo W, An Y, Li ZG, Luo SF, Sockalingam S, Lau CS, Mok MY, Lateef A, Franklyn K, Morton S, Navarra ST, Zamora L, Wu YJ, Hamijoyo L, Chan M, O'Neill S, Goldblatt F, Nikpour M, Morand EF; Asia-Pacific Lupus Collaboration. Association of the lupus low disease activity state (LLDAS) with health-related quality of life in a multinational prospective study. Arthritis Res Ther. 2017 Mar 20;19(1):62. doi: 10.1186/s13075-017-1256-6. PMID 28320433
- [Background] Golder V, Kandane-Rathnayake R, Hoi AY, Huq M, Louthrenoo W, An Y, Li ZG, Luo SF, Sockalingam S, Lau CS, Lee AL, Mok MY, Lateef A, Franklyn K, Morton S, Navarra ST, Zamora L, Wu YJ, Hamijoyo L, Chan M, O'Neill S, Goldblatt F, Morand EF, Nikpour M; Asia-Pacific Lupus Collaboration. Frequency and predictors of the lupus low disease activity state in a multi-national and multi-ethnic cohort. Arthritis Res Ther. 2016 Nov 9;18(1):260. doi: 10.1186/s13075-016-1163-2. PMID 27829463
- [Background] Franklyn K, Lau CS, Navarra SV, Louthrenoo W, Lateef A, Hamijoyo L, Wahono CS, Chen SL, Jin O, Morton S, Hoi A, Huq M, Nikpour M, Morand EF; Asia-Pacific Lupus Collaboration. Definition and initial validation of a Lupus Low Disease Activity State (LLDAS). Ann Rheum Dis. 2016 Sep;75(9):1615-21. doi: 10.1136/annrheumdis-2015-207726. Epub 2015 Oct 12. PMID 26458737
- [Background] Kandane-Rathnayake R, Golder V, Louthrenoo W, Luo SF, Jan Wu YJ, Li Z, An Y, Lateef A, Sockalingam S, Navarra SV, Zamora L, Hamijoyo L, Katsumata Y, Harigai M, Chan M, O'Neill S, Goldblatt F, Hao Y, Zhang Z, Al-Saleh J, Khamashta M, Takeuchi T, Tanaka Y, Bae SC, Lau CS, Hoi A, Nikpour M, Morand EF. Development of the Asia Pacific Lupus Collaboration cohort. Int J Rheum Dis. 2019 Mar;22(3):425-433. doi: 10.1111/1756-185X.13431. Epub 2018 Nov 5. PMID 30398013
- [Background] Golder V, Kandane-Rathnayake R, Huq M, Nim HT, Louthrenoo W, Luo SF, Wu YJ, Lateef A, Sockalingam S, Navarra SV, Zamora L, Hamijoyo L, Katsumata Y, Harigai M, Chan M, O'Neill S, Goldblatt F, Lau CS, Li ZG, Hoi A, Nikpour M, Morand EF; Asia-Pacific Lupus Collaboration. Lupus low disease activity state as a treatment endpoint for systemic lupus erythematosus: a prospective validation study. Lancet Rheumatol. 2019 Oct;1(2):e95-e102. doi: 10.1016/S2665-9913(19)30037-2. Epub 2019 Sep 6. PMID 38229349
- [Background] Golder V, Kandane-Rathnayake R, Huq M, Louthrenoo W, Luo SF, Wu YJ, Lateef A, Sockalingam S, Navarra SV, Zamora L, Hamijoyo L, Katsumata Y, Harigai M, Chan M, O'Neill S, Goldblatt F, Lau CS, Li ZG, Hoi A, Nikpour M, Morand EF; Asia Pacific Lupus Collaboration. Evaluation of remission definitions for systemic lupus erythematosus: a prospective cohort study. Lancet Rheumatol. 2019 Oct;1(2):e103-e110. doi: 10.1016/S2665-9913(19)30048-7. Epub 2019 Sep 25. PMID 38229337
- [Derived] Kandane-Rathnayake R, Zolio L, Choi J, Golder V, Louthrenoo W, Chen YH, Cho J, Lateef A, Hamijoyo L, Luo SF, Wu YJ, Navarra SV, Zamora L, Li Z, Sockalingam S, Katsumata Y, Harigai M, Hao Y, Zhang Z, Chan M, Kikuchi J, Takeuchi T, Oon S, Bae SC, Goldblatt F, O'Neill S, Ng KPL, Law A, Basnayake B, Tugnet N, Kumar S, Tee C, Tee M, Tanaka Y, Lau CS, Hoi A, Nikpour M, Morand EF. Predictors of damage accrual by organ domain in systemic lupus erythematosus. Rheumatology (Oxford). 2025 Nov 18:keaf610. doi: 10.1093/rheumatology/keaf610. Online ahead of print. PMID 41252474
- [Derived] Kandane-Rathnayake R, Hoi A, Louthrenoo W, Golder V, Chen YH, Cho J, Lateef A, Hamijoyo L, Luo SF, Wu YJ, Navarra S, Zamora L, Li Z, Yao H, Sockalingam S, Katsumata Y, Hao Y, Zhang Z, Basnayake BMDB, Chan M, Kikuchi J, Kaneko Y, Takeuchi T, Oon S, Bae SC, O'Neill S, Hassett G, Goldblatt F, Ng KPL, Poh YJ, Tugnet N, Sapsford M, Chan S, Tee C, Tee ML, Ohkubo N, Tanaka Y, Lau CS, Nikpour M, Morand E. Impact of glucocorticoid dose threshold in definition of lupus low disease activity state: a multinational observational cohort study. Lupus Sci Med. 2025 Nov 11;12(2):e001714. doi: 10.1136/lupus-2025-001714. PMID 41219118
- [Derived] Golder V, Kandane-Rathnayake R, Li N, Louthrenoo W, Chen YH, Cho J, Lateef A, Hamijoyo L, Luo SF, Wu YJ, Navarra SV, Zamora L, Li Z, Sockalingam S, Katsumata Y, Harigai M, Hao Y, Zhang Z, Basnayake D, Chan M, Kikuchi J, Takeuchi T, Bae SC, Goldblatt F, Oon S, O'Neill S, Ng K, Law A, Tugnet N, Kumar S, Tee C, Tee M, Ohkubo N, Tanaka Y, Lau CS, Hoi A, Nikpour M, Morand EF; Asia Pacific Lupus Collaboration. Association of sustained lupus low disease activity state with improved outcomes in systemic lupus erythematosus: a multinational prospective cohort study. Lancet Rheumatol. 2024 Aug;6(8):e528-e536. doi: 10.1016/S2665-9913(24)00121-8. Epub 2024 Jun 11. PMID 38876129
- [Derived] Golder V, Kandane-Rathnayake R, Louthrenoo W, Chen YH, Cho J, Lateef A, Hamijoyo L, Luo SF, Wu YJ, Navarra SV, Zamora L, Li Z, Sockalingam S, Katsumata Y, Harigai M, Hao Y, Zhang Z, Basnayake BMDB, Chan M, Kikuchi J, Takeuchi T, Bae SC, Oon S, O'Neill S, Goldblatt F, Ng KPL, Law A, Tugnet N, Kumar S, Tee C, Tee M, Ohkubo N, Tanaka Y, Lau CS, Nikpour M, Hoi A, Morand EF; Asia Pacific Lupus Collaboration. Comparison of Attainment and Protective Effects of Lupus Low Disease Activity State in Patients With Newly Diagnosed Versus Established Systemic Lupus Erythematosus. J Rheumatol. 2024 Aug 1;51(8):790-797. doi: 10.3899/jrheum.2023-0900. PMID 38490668
- [Derived] Kandane-Rathnayake R, Golder V, Louthrenoo W, Chen YH, Cho J, Lateef A, Hamijoyo L, Luo SF, Wu YJ, Navarra SV, Zamora L, Li Z, Sockalingam S, Katsumata Y, Harigai M, Hao Y, Zhang Z, Basnayake BMDB, Chan M, Kikuchi J, Takeuchi T, Bae SC, Oon S, O'Neill S, Goldblatt F, Ng KPL, Law A, Tugnet N, Kumar S, Tee C, Tee M, Ohkubo N, Tanaka Y, Yu D, Karyekar CS, Sing Lau C, Monk JA, Nikpour M, Hoi A, Morand EF; Asia-Pacific Lupus Collaboration. Lupus low disease activity state and remission and risk of mortality in patients with systemic lupus erythematosus: a prospective, multinational, longitudinal cohort study. Lancet Rheumatol. 2022 Dec;4(12):e822-e830. doi: 10.1016/S2665-9913(22)00304-6. Epub 2022 Oct 22. PMID 38261390
- See also: Related Info — http://www.asiapacificlupus.com/